CLINICAL TRIAL: NCT04168931
Title: Efficacy of Adding Trastuzumab to Standard Chemotherapy in Patients With Advanced HER2-negative Gastric Cancer and HER2 Positive Expression in Circulating Tumor Cells
Brief Title: Trastuzumab to Patients With Advanced Gastric Cancer With HER2 Positive Expression in CTC
Acronym: GASTHER2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment failure
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Rachel Riechelmann, Head of Clinical Oncology Department, AC Camargo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2793/19
Record Dates: First submitted 2019-11-05; First posted 2019-11-19 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Gastric Cancer Stage IV
Keywords: gastric cancer; HER2; trastuzumab; circulating tumor cells
MeSH Terms: conditions — Stomach Neoplasms; Neoplastic Cells, Circulating | interventions — Trastuzumab

STUDY DESIGN:
Intervention Model Description: This is a single-phase prospective unicentric phase II study evaluating HER2 expression in circulating tumor cells and their response to standard treatment with trastuzumab combination chemotherapy in cases of positive expression in patients with relapsed or metastatic gastric cancer with expression HER2 negative in the tumor tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Use of trastuzumab combination chemotherapy in patients with relapsed or metastatic gastric cancer with expression HER2 negative in the tumor tissue but positive in CTC.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — The first-line standard treatment for gastric cancer is based on fluoropyrimidine and platinum-containing chemotherapy (FOLFOX). When the tumor expresses HER2 3+ on IHC or 2+ and is confirmed by FISH, trastuzumab at the standard dose of 8 mg / kg in D1 of the first cycle is added, followed by 6 mg / kg every 2 weeks for the remaining cycles until disease progression, unacceptable toxicity. (3) We will use the same doses of trastuzumab, but HER2 positivity is determined by immunocytochemical expression and FISH in CTCs for patients with negative expression in tissue biopsy.
  Other Names: Experimental group

SUMMARY:
BACKGROUND: Gastric cancer is one of the most common cancers and is one of the most deadly cancers. Most patients have advanced disease and should receive first-line trastuzumab-associated chemotherapy when the biopsy is positive for immunocytochemical expression and / or HER2 gene amplification. A study conducted by our group noted that there may be disagreement in HER2 expression between circulating tumor cells (CTCs) and tumor tissue. However, the effectiveness of using anti-HER2 treatment when only CTC express HER2 is unknown. The present study aims to evaluate the expression of HER2 in patients with relapsed or metastatic gastric cancer and what would be the efficacy of adding trastuzumab to chemotherapy when tumor tissue is negative for HER2, but there is expression of this gene in CTCs.

OBJECTIVES: The primary objectives are to evaluate HER2 expression in circulating tumor cells of relapsed or metastatic gastric cancer patients with negative HER2 expression on tissue biopsy and response to standard treatment with combined anti-HER2 chemotherapy in this population. Secondary objectives are to assess the prognostic impact of HER2 positivity on circulating tumor cells in advanced gastric tumors and to evaluate HER2 expression in CTCs at the time of treatment progression.

METHODS: The investigators will prospectively evaluate HER2 expression in CTC and its response to treatment with standard chemotherapy and addition of trastuzumab in patients with relapsed or metastatic gastric cancer with positive expression of HER2 only in CTC. HER2 expression in tissue and in CTC will be evaluated by immunocytochemistry. Descriptive statistics will be used to report the results of categorical and continuous variables, and respective dispersion measures. Time-to-event variables will be reported in Kaplan Meyer medians and curves.

EXPECTED RESULTS: Upon completion of the study the investigators expect to show the frequency of HER2 expression in this specific population, higher radiological response rate with trastuzumab combination compared to chemotherapy alone, determine the prognostic impact associated with HER2 expression in CTCs and show the frequency of HER2 expression in CTCs at the time of study treatment progression. This study may open a new opportunity for anti-HER2 treatment for gastric cancer patients.

DETAILED DESCRIPTION:
INTRODUCTION Gastric cancer is one of the most common cancers worldwide. Its incidence varies according to its geographic region, being more common in East Asia, Eastern Europe and South America. About 70% of gastric neoplasms occur in developing countries. Globally, it is estimated that in 2018 over 1 million cases were diagnosed with about 780,000 deaths, making gastric cancer the 5th in frequency and 3rd in mortality. In Brazil, 13,540 new cases were diagnosed in 2018, being the third leading cause of cancer death in Brazil in males. Most patients already have inoperable, advanced or metastatic disease at diagnosis, thus requiring palliative treatment. Over 90% of stomach tumors are adenocarcinomas and, in terms of histology, Lauren's classification subdivided gastric cancer into diffuse (undifferentiated) or intestinal cancer and both types have distinct clinical and pathological features. The diffuse type occurs in all age groups with equal gender distribution, involves the body or the entire stomach and has a greater tendency to invade the gastric wall (resulting in plastic linitis) and to metastasize, as well as a faster disease progression and worse prognosis. On the other hand, the intestinal type predominates in men and the elderly, occurring predominantly in the gastric antrum and notch. Although both subtypes are related to H. pylori infection, in the intestinal type the evolution of sequential preneoplastic alterations is observed, namely: atrophic gastritis / intestinal metaplasia; dysplasia and adenocarcinoma. Such a sequence may not occur in diffuse type. There is also a rare genetically related type called hereditary diffuse gastric cancer (HDGC) that is not related to H. pylori infection. Diffuse-type adenocarcinoma is the major histological subtype of HDGC. In addition to diffuse hereditary gastric cancer syndrome, gastric cancer is present in the description of several other hereditary syndromes, such as Lynch syndrome, juvenile polyposis syndrome, Peutz-Jeghers syndrome, Familial Adenomatous Polyposis, ataxia-telangiectasia syndrome, Li-Fraumeni and Xeroderma Pigmentosa. Regardless of association with genetic syndrome or even histological type, it is necessary to investigate the amplification of the human epidermal growth factor 2 (HER2) gene in the case of recurrent or metastatic gastric cancer. Today of well-defined importance in gastric cancer, HER2 was initially recognized 30 years ago as an amplified oncogene in over 20% of breast cancers and, after the genomic revolution, has recently been seen to amplify in many other cancers. HER2 is a tyrosine kinase-like receptor that crosses the cell membrane of cells, with the extracellular half not coupling to ligands, but designed to recognize ligand-activated forms of family members as the factor of human epidermal growth (EGFR), HER3 or HER4, leading to dimerization with these receptors. The cytoplasmic part of HER2 and its partners contains a kinase domain that triggers HER2 kinase activity. The end result is phosphorylation at various tyrosine residues and recruitment of second messenger proteins for these phosphotyrosines. When the gene is amplified in cancer cells, the result is massive overexpression of HER2, which causes continuous activation of the various biological pathways that promote cell proliferation. For gastric cancer, positivity for HER2 expression, as assessed by immunohistochemistry (IHC) or in situ hybridization immunofluorescence (FISH), may vary between 8 and 36% between studies in the literature; However, those studies that considered only intestinal histology found positive expression of HER2 between 20 and 30% in patients' biopsies. A study conducted at AC Camargo identified 12% HER2 expression and 8% amplification in gastric tumors, with greater association with intestinal subtype and poor survival. Because it has a worse prognosis and has a target drug, treatment of tumors with HER2 amplification requires HER2-targeted agents, often in combination with chemotherapy or hormone therapies. Trastuzumab-associated chemotherapy (fluoro-uracil and platinum) is the first-line standard treatment for HER2-positive metastatic gastric cancer based on the phase III ToGA study (Trastuzumab for Gastric Cancer). This study recruited 594 patients and showed a median overall survival gain of 13.8 months for the combination versus 11.1 months in the chemotherapy arm alone (hazard ratio [HR], 0.74; 95% CI, 0.60 to 0.91; P = 0.0046). Survival gain was even more significant in the HER2 overexpressed subgroup (IHC 3+ or IHC 2+ with positive FISH), which achieved a median overall survival of 16 months. Regarding the second line, however, phase III studies failed to demonstrate the benefit of using anti-HER2 therapy. In the TyTan study, the addition of lapatinib in the second line was not superior to chemotherapy alone. In the GATSBY study, the use of trastuzumab emtansine was also not superior to taxane chemotherapy. In this study, 77% of patients received first-line anti-HER2 agents. Several clinical reasons may explain these disappointing results; One of these is resistance acquired after use of anti-HER2-based therapy. Another reason is the loss of HER2 expression, as reported in a study by Pietroantonio et al that demonstrated loss of HER2 positivity and overexpression in 32% of the tissue samples analyzed after anti-HER2 therapy. It is already known that in selective breast cancer treatment pressure can eradicate HER2-expressing clones and lead to proliferation of those HER2-negative clones, a phenomenon that can occur in gastric cancer because of the marked heterogeneity that exists in stomach tumors. In addition, it is known that HER2 expression discrepancy may exist between primary and metastatic or recurrent breast tumors (probably due to sample variability). In discordant cases, HER2-positive metastases from negative primary tumors are more frequent than the opposite. Therefore, it is recommended that metastatic disease on first relapse be biopsied as part of the investigation and HER2 status should be reevaluated. In cases of gastric cancer, this issue has not been widely explored.

In this sense, the GASTHER 1 study investigated the role of HER2 expression reassessment in stomach cancer at primary, metastatic or recurrent sites in patients whose primary tumor was initially negative for HER2 expression. The results showed a positive rescue of 8.7%, confirming the relevant heterogeneity of HER2 status. This heterogeneity, however, may also be associated with the HER2 status assessment method. A prospective study in patients with localized gastric adenocarcinoma and treated with perioperative chemotherapy at our institution found 69.4% agreement for HER2 expression in primary tumor tissue biopsy and in paired circulating tumor cells (CTCs). HER2 in CTCs showed higher positivity compared to tumor tissue (43% x 11%). The positivity in HER2 CTCs was 60% for HER2-negative localized gastric cancer patients treated with perioperative chemotherapy whose disease recurred. Also, HER2 expression in CTCs correlated with progression-free survival, but in the tumor tissue the same relationship was not found.

BACKGROUND Analysis of CTCs from the blood of patients with gastric adenocarcinoma may be useful to better understand the behavior of the disease, as well as patients more likely to respond to treatment, and may offer a less invasive way of investigating tumor dynamics. In addition, prospective evaluation of HER2 expression in CTCs has not been evaluated in metastatic gastric cancer, and the frequency with which this expression changes after first-line treatment with standard regimen with trastuzumab at the time of disease progression. Thus, this study is necessary to evaluate the frequency with which these phenomena occur and thus expand the knowledge of the dynamics of gastric cancer tumor biology.

Hypothesis:

Primary:

1. There is disagreement in HER2 expression positivity between diagnostic tissue biopsy (preferably metastasis) and circulating tumor cells in metastatic intestinal cancer.
2. Positivity for HER2 expression in circulating tumor cells in relapsed or metastatic gastric cancer may predict response to standard treatment with trastuzumab combination chemotherapy.

Secondary:

1. HER2 expression may have prognostic effect when positive in CTCs.
2. HER2 expression in CTCs may be modified following treatment with anti-HER2 therapy.

Objectives:

Primary:

1. Evaluate HER2 expression in circulating tumor cells of patients with relapsed or metastatic gastric cancer with negative HER2 expression on tissue biopsy.
2. To evaluate the response to standard treatment with combination chemotherapy with trastuzumab in relapsed or metastatic gastric cancer with positive expression of HER2 on CTC and negative on tissue biopsy.

Secondary:

1. To verify the prognostic impact of HER2 positivity in circulating tumor cells in advanced gastric tumors;
2. Evaluate HER2 expression in CTCs at the time of progression to standard first-line treatment with anti-HER2 therapy in patients who previously had HER2 positivity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Histological diagnosis of recurrent or metastatic gastric cancer
* Immunohistochemistry (IHC 0 or 1+) or FISH negative (if IHQ 2+) for HER2 on tissue biopsy, according to institutional routine
* Candidates to initiate first-line palliative treatment; Previous adjuvant treatment is allowed since its termination occurred at least 12 months ago
* ECOG performance range 0 to 2
* Informed consent form signed by patient or legal representative

Exclusion Criteria:

* Patients already on or previously using anti-HER2 therapy
* Left ventricular ejection fraction (LVEF) <55% baseline, as already evaluated in the gastric cancer routine
* Pregnant or lactating women
* Patients participating in other experimental drug protocols
* Patients who received previous palliative chemotherapy
* Another synchronic neoplasia requiring systemic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Radiological response rate | through study completion, an average of 5 years
  RECIST1.1 radiological response rate following standard treatment with combined chemotherapy with trastuzumab in relapsed or metastatic gastric cancer with positive expression of HER2 in CTC and negative in tumor tissue.
Frequency of HER2 expression | at screening before Day 1 Cycle 1 (each cycle is 14 days)
  Frequency of HER2 expression among circulating tumor cells of patients with relapsed or metastatic gastric cancer with negative expression of HER2 in tumor tissue
Frequency of HER2 expression | From date of randomization until the date of first documented progression, assessed up to 60 months
  Frequency of HER2 expression among circulating tumor cells of patients with relapsed or metastatic gastric cancer with negative expression of HER2 in tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Rachel SP Riechelmann, PhD, Principal Investigator — Head of Clinical Oncology Department
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Van Cutsem E, Bang YJ, Feng-Yi F, Xu JM, Lee KW, Jiao SC, Chong JL, Lopez-Sanchez RI, Price T, Gladkov O, Stoss O, Hill J, Ng V, Lehle M, Thomas M, Kiermaier A, Ruschoff J. HER2 screening data from ToGA: targeting HER2 in gastric and gastroesophageal junction cancer. Gastric Cancer. 2015 Jul;18(3):476-84. doi: 10.1007/s10120-014-0402-y. Epub 2014 Jul 20. PMID 25038874
- [Background] LAUREN P. THE TWO HISTOLOGICAL MAIN TYPES OF GASTRIC CARCINOMA: DIFFUSE AND SO-CALLED INTESTINAL-TYPE CARCINOMA. AN ATTEMPT AT A HISTO-CLINICAL CLASSIFICATION. Acta Pathol Microbiol Scand. 1965;64:31-49. doi: 10.1111/apm.1965.64.1.31. No abstract available. PMID 14320675
- [Background] Vauhkonen M, Vauhkonen H, Sipponen P. Pathology and molecular biology of gastric cancer. Best Pract Res Clin Gastroenterol. 2006;20(4):651-74. doi: 10.1016/j.bpg.2006.03.016. PMID 16997151
- [Background] Polkowski W, van Sandick JW, Offerhaus GJ, ten Kate FJ, Mulder J, Obertop H, van Lanschot JJ. Prognostic value of Lauren classification and c-erbB-2 oncogene overexpression in adenocarcinoma of the esophagus and gastroesophageal junction. Ann Surg Oncol. 1999 Apr-May;6(3):290-7. doi: 10.1007/s10434-999-0290-2. PMID 10340889
- [Background] Fitzgerald RC, Hardwick R, Huntsman D, Carneiro F, Guilford P, Blair V, Chung DC, Norton J, Ragunath K, Van Krieken JH, Dwerryhouse S, Caldas C; International Gastric Cancer Linkage Consortium. Hereditary diffuse gastric cancer: updated consensus guidelines for clinical management and directions for future research. J Med Genet. 2010 Jul;47(7):436-44. doi: 10.1136/jmg.2009.074237. PMID 20591882
- [Background] Lindor NM, McMaster ML, Lindor CJ, Greene MH; National Cancer Institute, Division of Cancer Prevention, Community Oncology and Prevention Trials Research Group. Concise handbook of familial cancer susceptibility syndromes - second edition. J Natl Cancer Inst Monogr. 2008;(38):1-93. doi: 10.1093/jncimonographs/lgn001. No abstract available. PMID 18559331
- [Background] Larsen Haidle J, MacFarland SP, Howe JR. Juvenile Polyposis Syndrome. 2003 May 13 [updated 2022 Feb 3]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1469/ PMID 20301642
- [Background] Hearle N, Schumacher V, Menko FH, Olschwang S, Boardman LA, Gille JJ, Keller JJ, Westerman AM, Scott RJ, Lim W, Trimbath JD, Giardiello FM, Gruber SB, Offerhaus GJ, de Rooij FW, Wilson JH, Hansmann A, Moslein G, Royer-Pokora B, Vogel T, Phillips RK, Spigelman AD, Houlston RS. Frequency and spectrum of cancers in the Peutz-Jeghers syndrome. Clin Cancer Res. 2006 May 15;12(10):3209-15. doi: 10.1158/1078-0432.CCR-06-0083. PMID 16707622
- [Background] Anaya DA, Chang GJ, Rodriguez-Bigas MA. Extracolonic manifestations of hereditary colorectal cancer syndromes. Clin Colon Rectal Surg. 2008 Nov;21(4):263-72. doi: 10.1055/s-0028-1089941. PMID 20011437
- [Background] Setia N, Clark JW, Duda DG, Hong TS, Kwak EL, Mullen JT, Lauwers GY. Familial Gastric Cancers. Oncologist. 2015 Dec;20(12):1365-77. doi: 10.1634/theoncologist.2015-0205. Epub 2015 Sep 30. PMID 26424758
- [Background] Ruiz-Saenz A, Moasser MM. Targeting HER2 by Combination Therapies. J Clin Oncol. 2018 Mar 10;36(8):808-811. doi: 10.1200/JCO.2017.77.1899. Epub 2018 Jan 30. No abstract available. PMID 29381433
- [Background] Boku N. HER2-positive gastric cancer. Gastric Cancer. 2014 Jan;17(1):1-12. doi: 10.1007/s10120-013-0252-z. Epub 2013 Apr 7. PMID 23563986
- [Background] Begnami MD, Fukuda E, Fregnani JH, Nonogaki S, Montagnini AL, da Costa WL Jr, Soares FA. Prognostic implications of altered human epidermal growth factor receptors (HERs) in gastric carcinomas: HER2 and HER3 are predictors of poor outcome. J Clin Oncol. 2011 Aug 1;29(22):3030-6. doi: 10.1200/JCO.2010.33.6313. Epub 2011 Jun 27. PMID 21709195
- [Background] Satoh T, Xu RH, Chung HC, Sun GP, Doi T, Xu JM, Tsuji A, Omuro Y, Li J, Wang JW, Miwa H, Qin SK, Chung IJ, Yeh KH, Feng JF, Mukaiyama A, Kobayashi M, Ohtsu A, Bang YJ. Lapatinib plus paclitaxel versus paclitaxel alone in the second-line treatment of HER2-amplified advanced gastric cancer in Asian populations: TyTAN--a randomized, phase III study. J Clin Oncol. 2014 Jul 1;32(19):2039-49. doi: 10.1200/JCO.2013.53.6136. Epub 2014 May 27. PMID 24868024
- [Background] Thuss-Patience PC, Shah MA, Ohtsu A, Van Cutsem E, Ajani JA, Castro H, Mansoor W, Chung HC, Bodoky G, Shitara K, Phillips GDL, van der Horst T, Harle-Yge ML, Althaus BL, Kang YK. Trastuzumab emtansine versus taxane use for previously treated HER2-positive locally advanced or metastatic gastric or gastro-oesophageal junction adenocarcinoma (GATSBY): an international randomised, open-label, adaptive, phase 2/3 study. Lancet Oncol. 2017 May;18(5):640-653. doi: 10.1016/S1470-2045(17)30111-0. Epub 2017 Mar 23. PMID 28343975
- [Background] Pietrantonio F, Caporale M, Morano F, Scartozzi M, Gloghini A, De Vita F, Giommoni E, Fornaro L, Aprile G, Melisi D, Berenato R, Mennitto A, Volpi CC, Laterza MM, Pusceddu V, Antonuzzo L, Vasile E, Ongaro E, Simionato F, de Braud F, Torri V, Di Bartolomeo M. HER2 loss in HER2-positive gastric or gastroesophageal cancer after trastuzumab therapy: Implication for further clinical research. Int J Cancer. 2016 Dec 15;139(12):2859-2864. doi: 10.1002/ijc.30408. Epub 2016 Sep 16. PMID 27578417
- [Background] Niikura N, Tomotaki A, Miyata H, Iwamoto T, Kawai M, Anan K, Hayashi N, Aogi K, Ishida T, Masuoka H, Iijima K, Masuda S, Tsugawa K, Kinoshita T, Nakamura S, Tokuda Y. Changes in tumor expression of HER2 and hormone receptors status after neoadjuvant chemotherapy in 21,755 patients from the Japanese breast cancer registry. Ann Oncol. 2016 Mar;27(3):480-7. doi: 10.1093/annonc/mdv611. Epub 2015 Dec 23. PMID 26704052
- [Background] Abrahao-Machado LF, Scapulatempo-Neto C. HER2 testing in gastric cancer: An update. World J Gastroenterol. 2016 May 21;22(19):4619-25. doi: 10.3748/wjg.v22.i19.4619. PMID 27217694
- [Background] Strien L, Leidenius M, von Smitten K, Heikkila P. Concordance between HER-2 and steroid hormone receptor expression between primary breast cancer, sentinel node metastases, and isolated tumor cells. Pathol Res Pract. 2010 Apr 15;206(4):253-8. doi: 10.1016/j.prp.2009.12.006. Epub 2010 Feb 6. PMID 20138441
- [Background] Wolff AC, Hammond ME, Hicks DG, Dowsett M, McShane LM, Allison KH, Allred DC, Bartlett JM, Bilous M, Fitzgibbons P, Hanna W, Jenkins RB, Mangu PB, Paik S, Perez EA, Press MF, Spears PA, Vance GH, Viale G, Hayes DF; American Society of Clinical Oncology; College of American Pathologists. Recommendations for human epidermal growth factor receptor 2 testing in breast cancer: American Society of Clinical Oncology/College of American Pathologists clinical practice guideline update. J Clin Oncol. 2013 Nov 1;31(31):3997-4013. doi: 10.1200/JCO.2013.50.9984. Epub 2013 Oct 7. PMID 24101045
- [Background] Park SR, Park YS, Ryu MH, Ryoo BY, Woo CG, Jung HY, Lee JH, Lee GH, Kang YK. Extra-gain of HER2-positive cases through HER2 reassessment in primary and metastatic sites in advanced gastric cancer with initially HER2-negative primary tumours: Results of GASTric cancer HER2 reassessment study 1 (GASTHER1). Eur J Cancer. 2016 Jan;53:42-50. doi: 10.1016/j.ejca.2015.09.018. Epub 2015 Dec 13. PMID 26693898
- [Background] Abdallah EA, Braun AC, Flores BCTCP, Senda L, Urvanegia AC, Calsavara V, Fonseca de Jesus VH, Almeida MFA, Begnami MD, Coimbra FJF, da Costa WL Jr, Nunes DN, Dias-Neto E, Chinen LTD. The Potential Clinical Implications of Circulating Tumor Cells and Circulating Tumor Microemboli in Gastric Cancer. Oncologist. 2019 Sep;24(9):e854-e863. doi: 10.1634/theoncologist.2018-0741. Epub 2019 Mar 7. PMID 30846515
- [Background] Voorzanger-Rousselot N, Garnero P. Biochemical markers in oncology. Part I: molecular basis. Part II: clinical uses. Cancer Treat Rev. 2007 May;33(3):230-83. doi: 10.1016/j.ctrv.2007.01.008. Epub 2007 Apr 11. PMID 17433551
- [Background] Mackey JR, Clemons M, Cote MA, Delgado D, Dent S, Paterson A, Provencher L, Sawyer MB, Verma S. Cardiac management during adjuvant trastuzumab therapy: recommendations of the Canadian Trastuzumab Working Group. Curr Oncol. 2008 Jan;15(1):24-35. doi: 10.3747/co.2008.199. PMID 18317582

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT04168931/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT04168931/ICF_000.pdf